CLINICAL TRIAL: NCT00000456
Title: Comparison of Cognitive Behavioral Therapy and Motivational Enhancement Therapy Plus Naltrexone for Alcoholism
Brief Title: Behavioral Therapy Plus Naltrexone for Alcoholism
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NIAAAANT09568; R01AA009568 (NIH)
Record Dates: First submitted 1999-11-02; First posted 1999-11-03 (Estimated); Last update posted 2010-10-04 (Estimated); Status verified 2010-10

CONDITIONS: Alcoholism; Alcohol Dependence
Keywords: Alcoholism; Alcohol Dependence; Naltrexone; Cognitive Behavioral Therapy
MeSH Terms: conditions — Alcoholism | interventions — Naltrexone; Cognitive Behavioral Therapy; Motivational Interviewing

INTERVENTIONS:
Drug: naltrexone (Revia)
Behavioral: cognitive behavior therapy
Behavioral: motivational enhancement therapy

SUMMARY:
This study will compare cognitive behavioral therapy with a time-limited motivational enhancement therapy to which naltrexone (Revia) or placebo medication is added. In this randomized clinical trial, 160 alcohol-dependent outpatients, after 5 days of abstinence, will receive one of the two psychosocial therapies and either naltrexone (Revia) or placebo for a 12-week treatment period. Abstinence rates, alcohol use, and time to alcohol relapse will be evaluated in all four groups along with measures of alcohol craving, biological measures of alcohol consumption, drinking consequences, changes in self-confidence for avoiding alcohol, and medication compliance. All study participants will be assessed for measures of outcome variables at 3 and 6 months after completing the treatment protocol.

ELIGIBILITY:
Inclusion Criteria:

* Meets criteria for alcohol dependence, has not had more than one previous inpatient medical detoxification.
* Consumes on average five standard drinks per day.
* Able to maintain sobriety for five days (with or without the aid of detoxification medications) as determined by self-report, collateral report, and breathalyzer measurements.
* Able to read and understand questionnaires and informed consent.
* Lives within 50 miles of the study site.

Exclusion Criteria:

* Currently meets criteria for any other psychoactive substance dependency disorder.
* Ever abused opiates.
* Used psychoactive substance abuse, except marijuana, within the last 30 days as evidenced by patient report, collateral report, and urine drug screen.
* Meets criteria for disorders of major depression, panic disorder, obsessive-compulsive disorder, post-traumatic stress syndrome, bipolar affective disorder, schizophrenia, or any other psychotic disorder or organic mental disorder.
* Meets criteria for dissociate disorder or eating disorders.
* Has current suicidal or homicidal ideation.
* Need for maintenance or acute treatment with any psychoactive medication including antiseizure medications.
* Current use of disulfiram (Antabuse).
* Clinically significant medical problems that would impair participation or limit medication ingestion.
* Hepatocellular disease.
* Sexually active females of child bearing potential who are pregnant, nursing, or who are not using a reliable form of birth control.
* Have current charges pending for a violent crime.
* Does not have a stable living situation and a reliable source of collateral reporting.
* Has taken an opiate antagonist drug in the last month.

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 1992-09; Primary Completion 2002-08 (Actual); Study Completion 2002-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ray Anton, MD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical Univ. of South Carolina, Charleston, South Carolina, United States

REFERENCES:
- [Result] Anton RF, Moak DH, Latham P, Waid LR, Myrick H, Voronin K, Thevos A, Wang W, Woolson R. Naltrexone combined with either cognitive behavioral or motivational enhancement therapy for alcohol dependence. J Clin Psychopharmacol. 2005 Aug;25(4):349-57. doi: 10.1097/01.jcp.0000172071.81258.04. PMID 16012278